CLINICAL TRIAL: NCT00169312
Title: The HMO Cancer Research Network (CRN) - Making Effective Nutritional Choices for Cancer Prevention: The MENU Study
Brief Title: Internet-Based Nutrition Education Program in Preventing Cancer in Participants of Health Maintenance Organizations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Josephine Ford Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Single
Other Study IDs: CDR0000514226; HFH-B40389
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Diet Therapy; Early Intervention, Educational

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Dietary Supplement: dietary intervention
Other: educational intervention
Other: internet-based intervention
Other: preventative dietary intervention
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Websites for nutrition education may be an effective method to help people eat more fruits and vegetables which may lower their risk of cancer.

PURPOSE: This randomized trial is studying how well an internet-based nutrition education program works in preventing cancer in participants of health maintenance organizations.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of internet-based nutrition education through untailored websites vs tailored websites (TW) vs TW and tailored human online behavioral interaction (HOBI) on the change in the number of daily fruit and vegetable servings consumed in participants of health maintenance organizations.

Secondary

* Compare the proportion of participants reporting consumption of 5 or more servings of fruits and vegetables per day at each 3-month interval.
* Compare the change in fruit and vegetable servings consumed from baseline to each intermediate time point.
* Compare the effects of intervention and observation time in these participants.
* Determine the effect of HOBI in these participants.
* Compare the impact of participant characteristics, in terms of the effect of the intervention on the change in fruit and vegetable intake, in these participants.

OUTLINE: This is a randomized, controlled, single-blind, multicenter study. Participants are stratified according to participating site, gender, and the participant's stage of change readiness. Participants are randomized to 1 of 3 intervention arms.

* Arm I (untailored websites): Participants are given unlimited access to an internet-based nutrition education program for up to 6 months. They are provided with 4 serial educational websites at 1, 3, 13, and 15 weeks after initial login. These internet sites provide general information about fruits and vegetables, new recipes with emphasis on fruits and vegetables, and how participants can incorporate them into their diet. Participants complete an online survey at 3 months.
* Arm II (tailored websites): Participants are given unlimited access to an internet-based nutrition education program for up to 6 months. They are provided with 4 serial educational websites, at the same timepoints as in arm I, with emphasis on vegetable consumption in weeks 1 and 13 and fruit consumption in weeks 3 and 15. Materials in these websites, including new recipes with emphasis on fruits and vegetables, are tailored and then revised (or retailored) based on individual health-risk information obtained at baseline and at the 3-month online survey.
* Arm III (tailored websites and human online behavioral interaction [HOBI]): Participants are given unlimited access to an internet-based nutrition education program for up to 6 months. Participants are provided with 4 serial educational websites with tailored materials as in arm II. They also receive HOBI (tailored e-mail messages) developed and then revised based on health-risk information obtained at baseline and the 3-month online survey.

In all arms, participants complete online surveys at 3, 6, and 12 months to measure fruit and vegetable intake and change in long-term risk behavior. For each survey, participants receive up to 6 automatically generated reminder e-mails and 1 mailed announcement.

PROJECTED ACCRUAL: A total of 2,619 participants were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current member of any of the following participating health maintenance organizations:

  * Group Health Cooperative
  * Kaiser Permanente, Colorado
  * Kaiser Permanante, Georgia
  * HealthPartners Research Foundation
  * Henry Ford Health System/Health Alliance Plan
* Must complete a web-based health survey prior to randomization

PATIENT CHARACTERISTICS:

* No medical or mental health condition that would be adversely affected by increased vegetable and fruit intake
* One participant allowed per household

PRIOR CONCURRENT THERAPY:

* No concurrent anticoagulation therapy (e.g., warfarin)
* No other concurrent medications that would be adversely affected by increased vegetable and fruit intake
* No grapefruit concurrently with any of the following medications:

  * Statin for high cholesterol
  * Blood pressure medications (e.g., Losartan)
  * Calcium channel blockers
  * Certain psychiatric medications (e.g., buspirone hydrochloride, triazolam [Halcion], carbamazepine, diazepam [Valium], or midazolam hydrochloride)
  * Immune suppressants (e.g., cyclosporine or tacrolimus)
  * Impotence medications (e.g., sildenafil [Viagra])
  * Methadone

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2619 (Estimated)
Dates: Start 2005-08; Study Completion 2007-06

PRIMARY OUTCOMES:
Change in the number of daily fruit and vegetable servings consumed from baseline to 12 months post intervention

SECONDARY OUTCOMES:
Change in the number of daily fruit and vegetable servings consumed at the 3- and 6-month post-intervention assessments
Proportion of participants who achieve an intake of 5 or more daily fruit and vegetable servings by 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Cole Johnson, PhD, Principal Investigator — Josephine Ford Cancer Center
Locations (4):
- United States (4):
  - Kaiser Permanente - Colorado, Denver, Colorado
  - Kaiser Permanente, Georgia, Atlanta, Georgia
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Group Health Cooperative, Seattle, Washington

REFERENCES:
- [Background] Stopponi MA, Alexander GL, McClure JB, Carroll NM, Divine GW, Calvi JH, Rolnick SJ, Strecher VJ, Johnson CC, Ritzwoller DP. Recruitment to a randomized web-based nutritional intervention trial: characteristics of participants compared to non-participants. J Med Internet Res. 2009 Aug 26;11(3):e38. doi: 10.2196/jmir.1086. PMID 19709990
- [Derived] Couper MP, Alexander GL, Zhang N, Little RJ, Maddy N, Nowak MA, McClure JB, Calvi JJ, Rolnick SJ, Stopponi MA, Cole Johnson C. Engagement and retention: measuring breadth and depth of participant use of an online intervention. J Med Internet Res. 2010 Nov 18;12(4):e52. doi: 10.2196/jmir.1430. PMID 21087922